CLINICAL TRIAL: NCT04609774
Title: Aerosol Transmission of Severe Acute Respiratory Syndrome Coronavirus: a Dilemma
Brief Title: Aerosol Transmission of Severe Acute Respiratory Syndrome Coronavirus of Coronavirus Disease 2019
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, VANINA LAURA PAGOTTO, principal investigator, Hospital Italiano de Buenos Aires
Other Study IDs: 1345
Record Dates: First submitted 2020-10-27; First posted 2020-10-30 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Coronavirus Disease (COVID-19)
Keywords: Severe Acute Respiratory Syndrome CoronaVirus 2; Airborne transmission
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Severe Acute Respiratory Syndrome CoronaVirus 2 detection — Severe Acute Respiratory Syndrome CoronaVirus 2 Detection by Real-Time Polymerase Chain Reaction and cell culture

SUMMARY:
There is little information on the characteristics of airborne severe acute respiratory syndrome coronavirus containing aerosols, their concentration, or their infectivity.The aim was to determine airborne severe acute respiratory syndrome coronavirus transmission, their infectivity in different areas such as patient's room and in medical staff área.

DETAILED DESCRIPTION:
The Corona Virus Disease 2019 is rapidly spreading throughout the world. Aerosol is a potential transmission route.

The transmission of severe acute respiratory syndrome coronavirus in humans is thought to be via at least 3 sources: 1) inhalation of liquid droplets produced by and/or 2) close contact with infected persons and 3) contact with surfaces contaminated with severe acute respiratory syndrome coronavirus. There are many respiratory diseases spread by the airborne route such as tuberculosis, measles and chickenpox. Several studies suggested that airborne spread may have played an important role in the transmission of that disease. At present, there is little information on the characteristics of airborne severe acute respiratory syndrome coronavirus containing aerosols, their concentration, or their infectivity.

The aim was to determine airborne severe acute respiratory syndrome coronavirus 2 transmission, their infectivity in in different areas such as patient's room and in medical staff area.

Methods

Cross sectional study of samples from environmental of patient´s room, and medical staff area. Samples will be taken of air using microbial air monitoring systems, and from different surfaces of patient's room and medical staff area, such as computers, mouse and personal protective equipment using cotton swabs. Viral RNA will be determined using Real-Time-Polymerase-Chain Reaction. In positive samples infectiveness will be determined by cell culture under biosecurity conditions.

Statistical analysis will be performed to determine prevalence of positive samples and positive cell culture whit STATA version 15.1.

informed consent will be obtained from all participants

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and more, with diagnoses of COVID-19 96 hours since the beginning of symptoms.
* Medical staff, nurses and/or physician taking care of patient whit COVID-19

Exclusion Criteria:

* Unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient and medical staff at Hospital Italiano de Buenos Aires
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Airborne transmission of Severe Acute Respiratory Syndrome CoronaVirus 2 | 9 moths
  Detection of Severe Acute Respiratory Syndrome CoronaVirus 2 RNA by Real Time Polymerase Chain Reaction and cell culture

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] To KK, Tsang OT, Yip CC, Chan KH, Wu TC, Chan JM, Leung WS, Chik TS, Choi CY, Kandamby DH, Lung DC, Tam AR, Poon RW, Fung AY, Hung IF, Cheng VC, Chan JF, Yuen KY. Consistent Detection of 2019 Novel Coronavirus in Saliva. Clin Infect Dis. 2020 Jul 28;71(15):841-843. doi: 10.1093/cid/ciaa149. PMID 32047895
- [Background] Shi F, Yu Q, Huang W, Tan C. 2019 Novel Coronavirus (COVID-19) Pneumonia with Hemoptysis as the Initial Symptom: CT and Clinical Features. Korean J Radiol. 2020 May;21(5):537-540. doi: 10.3348/kjr.2020.0181. Epub 2020 Mar 13. PMID 32174057
- [Background] Remuzzi A, Remuzzi G. COVID-19 and Italy: what next? Lancet. 2020 Apr 11;395(10231):1225-1228. doi: 10.1016/S0140-6736(20)30627-9. Epub 2020 Mar 13. PMID 32178769
- [Background] van Doremalen N, Bushmaker T, Morris DH, Holbrook MG, Gamble A, Williamson BN, Tamin A, Harcourt JL, Thornburg NJ, Gerber SI, Lloyd-Smith JO, de Wit E, Munster VJ. Aerosol and Surface Stability of SARS-CoV-2 as Compared with SARS-CoV-1. N Engl J Med. 2020 Apr 16;382(16):1564-1567. doi: 10.1056/NEJMc2004973. Epub 2020 Mar 17. No abstract available. PMID 32182409
- [Background] Chin AWH, Chu JTS, Perera MRA, Hui KPY, Yen HL, Chan MCW, Peiris M, Poon LLM. Stability of SARS-CoV-2 in different environmental conditions. Lancet Microbe. 2020 May;1(1):e10. doi: 10.1016/S2666-5247(20)30003-3. Epub 2020 Apr 2. No abstract available. PMID 32835322
- [Background] Liu Y, Ning Z, Chen Y, Guo M, Liu Y, Gali NK, Sun L, Duan Y, Cai J, Westerdahl D, Liu X, Xu K, Ho KF, Kan H, Fu Q, Lan K. Aerodynamic analysis of SARS-CoV-2 in two Wuhan hospitals. Nature. 2020 Jun;582(7813):557-560. doi: 10.1038/s41586-020-2271-3. Epub 2020 Apr 27. PMID 32340022
- [Background] Guo YR, Cao QD, Hong ZS, Tan YY, Chen SD, Jin HJ, Tan KS, Wang DY, Yan Y. The origin, transmission and clinical therapies on coronavirus disease 2019 (COVID-19) outbreak - an update on the status. Mil Med Res. 2020 Mar 13;7(1):11. doi: 10.1186/s40779-020-00240-0. PMID 32169119